CLINICAL TRIAL: NCT06572501
Title: Robot-assisted Laparoscopic Partial Nephrectomy Via the Extraperitoneal Approach in the Prone Position Versus the Lateral position-a Study Protocol for a Single-centre, Prospective, Randomised Controlled Trial
Brief Title: Robot-assisted Laparoscopic Partial Nephrectomy Via the Extraperitoneal Approach in the Prone Position Versus the Lateral Position
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-SR-614.A1
Record Dates: First submitted 2024-08-04; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Renal Tumor; Prone Position; Robotic Assisted Partial Nephrectomy
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prone position (Experimental): Robot-assisted laparoscopic partial nephrectomy via extraperitoneal approach in the prone position
  Interventions: Procedure: Robot-assisted laparoscopic partial nephrectomy via extraperitoneal approach in the prone position
- Lateral position (Active Comparator): Robot-assisted laparoscopic partial nephrectomy via extraperitoneal approach in the lateral position
  Interventions: Procedure: Robot-assisted laparoscopic partial nephrectomy via extraperitoneal approach in the lateral position

INTERVENTIONS:
Procedure: Robot-assisted laparoscopic partial nephrectomy via extraperitoneal approach in the prone position — This group of patients underwent robotic-assisted laparoscopic partial nephrectomy via extraperitoneal approach in the prone position
  Arms: Prone position
Procedure: Robot-assisted laparoscopic partial nephrectomy via extraperitoneal approach in the lateral position — This group of patients underwent robotic-assisted laparoscopic partial nephrectomy via extraperitoneal approach in the lateral position
  Arms: Lateral position

SUMMARY:
The goal of this clinical trial is to investigate whether robot-assisted laparoscopic partial nephrectomy by extraperitoneal approach in the prone position had any advantages over the traditional lateral position. The main questions it aims to answer are:

Is prone surgery safe and feasible, and what are the advantages over the traditional lateral position? Does surgery in the prone position have an impact on the patients' prognosis? Researchers will compare prone position to lateral position to see if robot-assisted laparoscopic partial nephrectomy by extraperitoneal approach in the prone position has any advantages over the traditional lateral position and whether it has any significant effect on the prognosis of the patients.

Participants will be randomly allocated 1:1 to two groups: prone position group and lateral position group. The enrolled patients will be underwent robotic-assisted laparoscopic partial nephrectomy via extraperitoneal approach according to the corresponding positions of their groups. Demographic indicators and perioperative-related indicators will be counted and recorded. CT or MRI and related biochemical examinations will be reviewed at 1 month, 3 months, 6 months and 1 year after surgery, and every 1 year thereafter. The similarities and differences of the indicators in different positions will be analysed, and subgroup analyses will be performed according to the corresponding results.

ELIGIBILITY:
Inclusion Criteria:

1. . Patients with preoperative imaging suggestive of renal occupancy;
2. . Sex is not limited;
3. . Age ≥18 years;
4. . Clinical staging consistent with indications for partial nephrectomy;
5. . Suitable for robotic-assisted laparoscopic partial nephrectomy via extraperitoneal approach as judged by relevant preoperative clinical data;
6. . Agree to provide basic clinical information and pathological and imaging data for scientific research and sign an informed consent form;
7. . Agree to provide monitoring results during the follow-up recurrence monitoring process.

Exclusion Criteria:

1. . Patients who did not meet the indications for partial nephrectomy and did not undergo robotic-assisted laparoscopic partial nephrectomy via extraperitoneal approach;
2. . Patients who refuse to undergo or cannot tolerate surgery in the appropriate position;
3. . Patients with incomplete documentation of relevant data to provide accurate demographic, perioperative, and prognostic data;
4. . Any condition which, in the opinion of the investigator, may be detrimental to the subject or result in the inability of the subject to meet or perform the requirements of the study;
5. . Patients who are unable to provide written informed consent;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-08-06 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Tumour characteristics checklist | Baseline ( before surgery)
  We will record tumor size (cm), location, position, laterality through preoperative imaging.
Tumour characteristics assessed by RENAL nephrometry score | Baseline ( before surgery)
  The R.E.N.A.L. Nephrometry Score consists of (R)adius (tumor size as maximal diameter), (E)xophytic/endophytic properties of the tumor, (N)earness of tumor deepest portion to the collecting system or sinus, (A)nterior (a)/posterior (p) descriptor and the (L)ocation relative to the polar line. The suffix h (hilar) is assigned to tumors that abut the main renal artery or vein. Of the 5 components 4 are scored on a 1, 2 or 3-point scale with the 5th indicating the anterior or posterior location of the mass relative to the coronal plane of the kidney. Higher scores indicate more complex tumour.
Demographics of patients | Baseline ( before surgery)
  age (year)
Demographics of patients | Baseline ( before surgery)
  gender
Demographics of patients | Baseline ( before surgery)
  BMI (kg/m2)
Demographics of patients | Baseline ( before surgery)
  American Society of Anesthesiology score
Demographics of patients | Baseline ( before surgery)
  age-adjusted charlson comorbidity index
Demographics of patients | Baseline ( before surgery)
  preoperative estimated glomerular filtration rate(ml/min/1.73m2).
Perioperative data | Intraoperative status
  intraoperative average PaCO2(mmHg).
Perioperative data | Intraoperative status
  operation time(minute)
Perioperative data | Intraoperative status
  hilar access time(minute)
Perioperative data | Intraoperative status
  warm ischemia time(minute).
Perioperative data | Intraoperative status
  suturing time(minute).
Perioperative data | Intraoperative status
  estimated blood loss(ml).
Perioperative data | Intraoperative status
  transfusion rate(%)
Perioperative data | Intraoperative status
  rate of positive surgical margin(%)
Perioperative data | Intraoperative status
  conversion rates to open surgery(%)
Perioperative data | Intraoperative status
  conversion rates to radical nephrectomy(%)
Perioperative data | Intraoperative status
  reoperation rate(%)
Perioperative data | Postoperative 30 days
  postoperative length of stay (day).
postoperative data | Postoperative 3/30/60/90 days and 1/2/3 years
  postoperative estimated glomerular filtration rate(ml/min/1.73m2).
Incidence of postoperative complications | Postoperative 3/30/60/90 days and 1/2/3 years
  We will assess the complications by conducting telephone follow-up, as well as reviewing the results of postoperative radiological and laboratory tests. The complications included whether the patients experienced bleeding, infection, urinary fistula and renal insufficiency.
Tumour recurrence or metastasis | Postoperative 30/60/90 days and 1/2/3 years
  We will conduct telephone follow-up and review the results of postoperative radiological tests to see whether tumour recurrence or metastasis occurred.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China